CLINICAL TRIAL: NCT02596737
Title: WittyFit - Live Your Work Differently
Acronym: WittyFit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: WittyFit (Industry); Australian Catholic University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CHU-0247
Record Dates: First submitted 2015-10-15; First posted 2015-11-04 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-11

CONDITIONS: Mortality
Keywords: health; work; lifestyle; behavior; management; stress; physical activity; nutrition; mortality; morbidity; public health
MeSH Terms: conditions — Behavior; Motor Activity

ARMS (1):
- workers (Other): Workers will fulfil a visual analog scale of Well-being regarding 3 main categories: "Physically", "Mentally", "At Work".
  Interventions: Behavioral: wittyFit concept

INTERVENTIONS:
Behavioral: wittyFit concept

SUMMARY:
Individuals spend one third of their life working. Age of retirement is regularly pushed back. The main challenge in the nearest future will be to maintain workers health to deal with their work till retirement. Morbidity before retirement has a huge cost, both in public health and economically for companies. Numerous factors increase morbidity such as stress at work, sedentary and low physical activity, and poor nutrition habits. Nowadays, digital world wildly invades lives and offer a no-limit possibility to interact with individuals, everywhere. Thus, a software able to understand an individual in its globality seems to address this challenge. Moreover, managers need to understand the actions needed within their company. The objective of WittyFit is to increase life expectancy and well-being. WittyFit will constitute a powerful database to build strong evidence and new knowledge on the relationships between work, behavior, and health, based on a large amount of epidemiological data.

DETAILED DESCRIPTION:
1. Whereas other interventional software focus on a specific aim (relaxation, musculo-skeletal disorder, etc), Wittyfit has the ambition to promote health with a global understanding of workers, based on continuous and updated scientific knowledge (evidence based medicine). A feedback is given on targets screened from questionnaires through e-learning and personalized motivating messages.
2. The second novelty of WittyFit is that managers will also have an anonymous feedback on the general state of health and problems encountered by its employees, in general or by department if the sample size is sufficiently high. Managers will indeed be able to target specific actions such as promoting physical activity at work or helping its employees to quit smoking.
3. Third, WittyFit is a prevention tool in collaboration with occupational medicine, which may help to detect a high risk toward the integrity of an employee.
4. Moreover, WittyFit is in fact based on two databases: "WittyFit" which deals with behavioral data, and "WittyFit Research" which deals with medical data. To guarantee the highest level of security, the two databases are separate and do not communicate together; physicians from the CHU of Clermont-Ferrand will be the only individuals with an access to medical data.
5. When a worker will leave Wittyfit, the company will encode three possibilities: retirement, move for another company, or premature death. Therefore, WittyFit will have the ability to have mortality as a primary outcome.
6. Finally, WittyFit may constitute a powerful database to build strong evidence and new knowledge on the relationships between lifestyle and health, based on huge amount of epidemiological data.
7. At last, WittyFit will evolve with the waves of connected objects further increasing its data accuracy, with the use of devices such as pedometers, heart rate monitors, accelerometers, thermometer, etc.
8. WittyFit is building a rainbow: work (shiftwork, sedentary job, particular occupations, etc) / psychology and physiology / statistics modeling / public health, and in general, health.

ELIGIBILITY:
Inclusion Criteria:

* All workers who want to participate to the WittyFit concept will be included.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-05; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | every year, up to 10 years
  When a worker will leave Wittyfit, the company will encode three possibilities: retirement, move for another company, or premature death.

SECONDARY OUTCOMES:
visual analog scale of physical well-being | every 15 days, up to 10 years
  However individuals will be able to spontaneously complete this data more frequently
visual analog scale of mental well-being | every 15 days, up to 10 years
  however individuals will be able to spontaneously complete this data more frequently
visual analog scale of well-being at-work | every 15 days, up to 10 years
  however individuals will be able to spontaneously complete this data more frequently
Nutritional intake measured by questionnaire | every 6 months, up to 10 years
  however individuals will be able to spontaneously complete this data more frequently
Physical activity measured by questionnaire | every 6 months, up to 10 years
  however individuals will be able to spontaneously complete this data more frequently
Sleep measured by questionnaire | every 6 months, up to 10 years
  however individuals will be able to spontaneously complete this data more frequently
Musculo-skeletal disorders measured by questionnaire | every 6 months, up to 10 years
  Every participant can fulfil questionnaires when he wants. however individuals will be able to spontaneously complete this data more frequently
Hospital and Anxiety Depression Scale | every 6 months, up to 10 years
  however individuals will be able to spontaneously complete this data more frequently
Stress and Mood measured by questionnaire | every 6 months, up to 10 years
  however individuals will be able to spontaneously complete this data more frequently
job strain measured by questionnaire | every 6 months, up to 10 years
  however individuals will be able to spontaneously complete this data more frequently
latitude decision measured by questionnaire | every 6 months, up to 10 years
  however individuals will be able to spontaneously complete this data more frequently
work organization and tasks measured by questionnaire | every 6 months, up to 10 years
  however individuals will be able to spontaneously complete this data more frequently
social support measured by questionnaire | every 6 months, up to 10 years
  however individuals will be able to spontaneously complete this data more frequently
recognition measured by questionnaire | every 6 months, up to 10 years
  however individuals will be able to spontaneously complete this data more frequently
disease and medical history measured by questionnaire | every 12 months, up to 10 years
routine medications measured by questionnaire | every 12 months, up to 10 years
number of days of sick leave provided by the employer | every 12 months, up to 10 years
sales turnover of the company, provided by the employer | every 12 months, up to 10 years
net income or net gain of the company, provided by the employer | every 12 months, up to 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Colin-Chevalier R, Pereira B, Dewavrin S, Cornet T, Baker JS, Dutheil F. Psychosocial well-being index and sick leave in the workplace: a structural equation modeling of Wittyfit data. Front Psychol. 2025 Jan 24;16:1385708. doi: 10.3389/fpsyg.2025.1385708. eCollection 2025. PMID 39927216
- [Derived] Dutheil F, Palgen C, Brousse G, Cornet T, Mermillod M, Lakbar I, Vallet G, Baker JS, Schmidt J, Charbotel B, Pereira B, Delamarre L. Validation of visual analog scales of mood and anxiety at the workplace. PLoS One. 2024 Dec 31;19(12):e0316159. doi: 10.1371/journal.pone.0316159. eCollection 2024. PMID 39739967
- [Derived] Colin-Chevalier R, Dutheil F, Benson AC, Dewavrin S, Cornet T, Lambert C, Pereira B. Stress and job satisfaction over time, the influence of the managerial position: A bivariate longitudinal modelling of Wittyfit data. PLoS One. 2024 Mar 4;19(3):e0298126. doi: 10.1371/journal.pone.0298126. eCollection 2024. PMID 38437204
- [Derived] Colin-Chevalier R, Pereira B, Dewavrin S, Cornet T, Zak M, Benson AC, Dutheil F. The Managerial Role and Psychosocial Factors of Job Satisfaction: A Cross-sectional Study Among Wittyfit's Users. J Occup Environ Med. 2024 Feb 1;66(2):e61-e67. doi: 10.1097/JOM.0000000000003017. Epub 2023 Nov 15. PMID 38013387
- [Derived] Dutheil F, Pereira B, Bouillon-Minois JB, Clinchamps M, Brousses G, Dewavrin S, Cornet T, Mermillod M, Mondillon L, Baker JS, Schmidt J, Moustafa F, Lanhers C. Validation of Visual Analogue Scales of job demand and job control at the workplace: a cross-sectional study. BMJ Open. 2022 Mar 17;12(3):e046403. doi: 10.1136/bmjopen-2020-046403. PMID 35301199
- [Derived] Colin-Chevalier R, Pereira B, Benson AC, Dewavrin S, Cornet T, Dutheil F. The Protective Role of Job Control/Autonomy on Mental Strain of Managers: A Cross-Sectional Study among Wittyfit's Users. Int J Environ Res Public Health. 2022 Feb 14;19(4):2153. doi: 10.3390/ijerph19042153. PMID 35206335
- [Derived] Serole C, Auclair C, Prunet D, Charkhabi M, Lesage FX, Baker JS, Mermillod M, Gerbaud L, Dutheil F. The Forgotten Health-Care Occupations at Risk of Burnout-A Burnout, Job Demand-Control-Support, and Effort-Reward Imbalance Survey. J Occup Environ Med. 2021 Jul 1;63(7):e416-e425. doi: 10.1097/JOM.0000000000002235. PMID 34184659
- [Derived] Clinchamps M, Auclair C, Prunet D, Pfabigan D, Lesage FX, Baker JS, Parreira L, Mermillod M, Gerbaud L, Dutheil F. Burnout Among Hospital Non-Healthcare Staff: Influence of Job Demand-Control-Support, and Effort-Reward Imbalance. J Occup Environ Med. 2021 Jan 1;63(1):e13-e20. doi: 10.1097/JOM.0000000000002072. PMID 33149005
- [Derived] Dutheil F, Duclos M, Naughton G, Dewavrin S, Cornet T, Huguet P, Chatard JC, Pereira B. WittyFit-Live Your Work Differently: Study Protocol for a Workplace-Delivered Health Promotion. JMIR Res Protoc. 2017 Apr 13;6(4):e58. doi: 10.2196/resprot.6267. PMID 28408363